CLINICAL TRIAL: NCT07038447
Title: A Phase 1 Open-label, Multiregional, Multicenter, Basket Study Evaluating the Safety and Efficacy of KITE-363, an Autologous Anti-CD19/CD20 CAR T-cell Therapy in Participants With Refractory Autoimmune Diseases
Brief Title: A Study of KITE-363 in Participants With Refractory Autoimmune Diseases
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-720-0203
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis; Systemic Sclerosis; Idiopathic Inflammatory Myopathy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Scleroderma, Systemic; Myositis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: KITE-363 (Dose Escalation) (Experimental): Participants with refractory autoimmune diseases will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by 2 dose escalations of KITE-363 chimeric antigen receptor (CAR) transduced autologous T cells to find the Phase 1b recommended dose.
  Interventions: Biological: KITE-363; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1b: KITE-363 (Dose Expansion) (Experimental): Participants with refractory autoimmune diseases will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed Phase 1ab recommended dose of KITE-363 CAR T cells.
  Interventions: Biological: KITE-363; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: KITE-363 — A single infusion of CAR-transduced autologous T cells administered intravenously
Drug: Fludarabine — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously

SUMMARY:
This study will have two Phases: Phase 1a and Phase 1b. The goal of this clinical study is to learn more about the study drug KITE-363, to establish dosing, tolerability, safety, and preliminary efficacy of KITE-363 in participants with refractory autoimmune diseases.

The primary objectives of this study are:

Phase 1a: To evaluate the safety and tolerability of KITE-363 in participants with autoimmune disease. To determine the recommended dose for Phase 1b.

Phase 1b: To evaluate the safety and efficacy of KITE-363 in participants with autoimmune disease.

ELIGIBILITY:
Key Inclusion Criteria:

Inclusion Criteria for systemic lupus erythematosus (SLE) and lupus nephritis (LN):

* Age ≥ 18 and ≤ 75 years
* Meet the European Alliance of Associations for Rheumatology (EULAR)- American College of Rheumatology (ACR) 2019 classification criteria for SLE
* Presence of either double-stranded deoxyribonucleic acid (DNA) anti- double-stranded DNA (anti-dsDNA) and/or anti-Smith antibodies at screening per local laboratory.
* Moderate to severe, active disease defined as at least one British Isles Lupus Assessment Group (BILAG-A) score or 2 BILAG B (excluding constitutional and/or neuropsychiatric organ system).
* Refractory to steroids and inadequate response or intolerance to at least 2 of the following treatments, used for at least 3 months each: cyclophosphamide, mycophenolate mofetil or its derivatives, belimumab, anifrolumab, rituximab, obinutuzumab, methotrexate, azathioprine, cyclosporin, tacrolimus, or voclosporin.
* For LN: Refractory to steroids and inadequate response or intolerance to at least 2 of the following treatments, used for at least 3 months each: cyclophosphamide, mycophenolate mofetil or its derivatives, belimumab, rituximab, obinutuzumab, azathioprine, cyclosporin, tacrolimus, or voclosporin

Inclusion Criteria for LN:

* Renal biopsy-proven Class III or intravenous (IV) ± V LN according to the revised International Society of Nephrology and Renal Pathology Society (ISN/RPS) criteria within 6 months prior to or during screening
* Evidence of active LN at screening

Inclusion Criteria for systemic sclerosis (SSc):

* Age ≥ 18 and ≤ 60 years
* Early systemic sclerosis according to ACR/EULAR 2013 classification criteria with active skin disease and/or progressive ILD
* Refractory or intolerance to 1 of the following for a minimum of 3 months and/or contraindication: mycophenolate mofetil or its derivatives, methotrexate, tocilizumab (or other IL-6 inhibitor), rituximab (or other B-cell depleting agent), nintedanib (or other antifibrotic agents), cyclophosphamide.
* High-resolution computer tomography (HRCT) scan and pulmonary function test (PFT) within 3 months prior to screening to evaluate for presence of SSc-ILD.

Inclusion Criteria for idiopathic inflammatory myopathy (IIM):

* Age ≥ 18 years
* IIM based on EULAR/ACR 2017 classification (excluding inclusion body myositis).
* Active disease demonstrated by electromyography (EMG). Magnetic resonance imaging (MRI) or muscle enzyme
* Moderate to severe disease activity
* Positive for myositis specific antibodies for patients with non-dermatomyostitis IIM
* HRCT scan and PFT within 3 months prior to screening to evaluate for presence of IIM-ILD.
* Refractory or intolerance to at least 1 month of glucocorticoids and standardized use of at least 2 immunosuppressant/modulator (eg, intravenous gamma globulins, methotrexate, mycophenolate mofetil and its derivatives, azathioprine, cyclophosphamide, calcineurin inhibitors, Janus kinase (JAK) inhibitors, rituximab or other B-cell depleting agent).

Inclusion Criteria for all Cohorts:

* Adequate hepatic, renal, pulmonary, and cardiac function.

Key Exclusion Criteria:

Exclusion Criteria for all Cohorts:

* Females of childbearing potential who are pregnant or breast feeding.
* Dialysis within the past year.
* History of malignancy, within the last 5 years.
* Hypogammaglobulinemia requiring immunoglobulin replacement.
* History of autologous or allogeneic stem cell transplant and/or organ transplant.
* Prior treatment with cellular therapy, gene therapy and/or T-cell engager therapy.
* Known history of HIV infection, or hepatitis B or C virus infections.
* Active or untreated latent tuberculosis (TB).
* Active or uncontrolled infections.
* Nonspecific, overlap, mixed autoimmune diseases not clearly identified into any of the studied cohorts.

Exclusion Criteria for LN:

* Significant pre-existing damage or rapidly progressive glomerulonephritis (GN).

Exclusion Criteria for SLE:

* Drug-induced SLE.
* Catastrophic antiphospholipid syndrome.
* Thrombotic thrombocytopenic purpura.
* Active or unstable lupus neuropsychiatric manifestations within last 6 months.

Exclusion Criteria for SSc:

* Digital ulceration or necrosis with infection.
* Severe pulmonary hypertension.
* History of systemic sclerosis renal crisis within 12 months prior to enrollment.
* History of active bleeding related to gastric antral vascular ectasia.

Exclusion Criteria for IIM:

* Other inflammatory and noninflammatory myopathies.
* Severe, irreversible muscle damage.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants Experiencing Adverse Events Defined as Dose-limiting Toxicities (DLTs) After the Infusion of KITE-363 | Up to 2 years
Phase 1b: All Cohorts Percentage of Participants Experiencing Treatment-emergent Adverse Event (TEAEs) | Up to 2 years
Phase 1b: Systemic lupus erythematosus (SLE)/ Lupus Nephritis (LN): Proportion of Participants Meeting DORIS Remission and Lupus low Disease Activity State (LLDAS) Criteria at Month 6 | Month 6
Phase 1b: Lupus Nephritis (LN): Proportion of Participants Achieving a Complete Renal Response | Month 6
Phase 1b: Systemic Sclerosis (SSc) Cohort: Proportion of Participants with Improvement in Disease Activity by the Revised Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (rCRISS) at Month 6 | Month 6
Phase 1b: Systemic Sclerosis (SSc) Cohort: Proportion of Participants With Progressive Interstitial Lung Disease (ILD), no Worsening of Pulmonary Function at Month 6 | Month 6
Phase 1b: Idiopathic Inflammatory Myopathy: Proportions of Participants Meeting European League Against Rheumatism (EULAR)-American College of Rheumatology (ACR) Moderate and Major response 2016 Criteria in Total Improvement Score (TIS) at Month 6 | Month 6

SECONDARY OUTCOMES:
Characterization of Product, Including T-cell Phenotype as Assessed by Percent Change From Baseline in cluster of differentiation 3 (CD3)+ Cells and T Cells | Baseline up to 2 years
Pharmacokinetic parameter: Serum Concentration of KITE-363 CAR T-cells | Up to 2 years
Pharmacokinetic parameter: Peak Concentration (Cmax) for KITE-363 CAR T-cells | Up to 2 years
Pharmacokinetic parameter: AUC for KITE-363 CAR T-cells | Up to 2 years
  AUC is defined as the area under the concentration time curve for KITE-363 CAR T-cells.
Pharmacokinetic parameter: Time to Peak Serum Concentration (Tmax) for KITE-363 CAR T-cells | Up to 2 years
Pharmacodynamic Parameters: Serum Concentration of Pro-inflammatory and Immune-modulating Cytokines, Chemokines, and Effector molecules, Autoantibodies, Muscle Enzymes, and Complement factors in blood over time | Up to 2 years
Pharmacodynamic Parameters: Peak Serum Concentration (Cmax) for Pro-inflammatory and Immune-modulating Cytokines, Chemokines, and Effector molecules, Autoantibodies, Muscle Enzymes, and Complement factors | Up to 2 years
Pharmacodynamic Parameters: AUC for Pro-inflammatory and Immune-modulating Cytokines, Chemokines, and Effector molecules, Autoantibodies, Muscle Enzymes, and Complement factors | Up to 2 years
  AUC is defined as the area under the concentration time curve.
Pharmacodynamic Parameters: Time to Peak Serum Concentration (Tmax) for Pro-inflammatory and Immune-modulating Cytokines, Chemokines, and Effector molecules, Autoantibodies, Muscle Enzymes, and Complement factors | Up to 2 years
Percentage of Participants with Antibodies Against KITE-363 CAR T cells | Up to 2 years
Change from Baseline in Levels of B cells | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (5):
- United States (2):
  - City of Hope, Duarte, California
  - Stanford University, Stanford, California
- Australia (2):
  - Concord Repatriation General Hospital, Syndey, New South Wales
  - St Vincent's Hospital, Fitzroy, Victoria
- Jewish General Hospital, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07038447